CLINICAL TRIAL: NCT02843412
Title: The Clinical Study of Assessing HER-2 Expression in Gastric Cancer With Extra Tumor Tissue Paraffin Blocks Using Immunohistochemistry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 123
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Gastric Cancer Surgical Specimens,18-80 Years Old, at Least Two Tumor Tissue Blocks
Keywords: Gastric cancer; Her2/neu; Dual paraffin blocks; Trastuzumab; Clinical Prospective Multicenter Cohort Study
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- group 1: choose one tumor tissue paraffin blocks
- group 2: choose two tumor tissue paraffin blocks
  Interventions: Procedure: choose two tumor tissue paraffin blocks

INTERVENTIONS:
Procedure: choose two tumor tissue paraffin blocks
  Groups: group 2

SUMMARY:
Background: Gastric cancer (GC) is major global health concern and the second leading cause of cancer deaths worldwide. Amplification of Her2/neu gene and/or overexpression of the Her2/neu protein have been observed in GC. Trastuzumab (Herceptin™) is an anti-Her2/neu antibody, which has been successfully applied in GC. However, the intratumoral heterogeneity of Her2/neu overexpression and amplification in GC should be noticed. The investigators investigated the significance of evaluating Her2/neu expression in different paraffin blocks of tumor tissue in GC.

Methods: 2000 GC patients from ten centers, patients were divided into a cohort using one tumor tissue paraffin block (cohort 1, n=1000) and a cohort using dual tumor tissue paraffin blocks (cohort 2, n=1000) when evaluating Her2/neu expression status by immunohistochemistry (IHC). In cohort 2, the investigators combined the results from two different paraffin blocks and used the higher one as the final score.

ELIGIBILITY:
Inclusion Criteria:

* Undergone curative surgery of gastric cancer,
* 18-80 years old.

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Undergone curative surgery of gastric cancer, 18-80 years old
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
compare the positive rate | 3 years

REFERENCES:
- [Derived] Xu C, Sun M, Jin M, Li Z, Qin R, Ren G, Sun W, Chen L, Luan L, Liu Y, Jiang D, Chen L, Luo R, Hou Y. Dual block HER2 assessment increased HER2 immunohistochemistry positive rate in resected specimens of gastric cancer: a prospective multicenter clinical trial from China. Diagn Pathol. 2022 Jun 28;17(1):54. doi: 10.1186/s13000-022-01230-7. PMID 35765007